CLINICAL TRIAL: NCT04327193
Title: The Effectiveness of Driving Pressure Based Ventilation Strategy in Robot-assisted Laparoscopic Surgeries With Steep Trendelenburg Position: a Randomized Controlled Trial
Brief Title: Driving Pressure-guided PEEP Titration in Robot-assisted Laparoscopic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Susie Yoon, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SYoon_DP_RALP
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Atelectasis, Postoperative Pulmonary
Keywords: Driving pressure; Positive end-expiratory pressure; Lung ultrasound
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving pressure (Experimental): The selected PEEP which makes the driving pressure lowest is applied during the operation.
  Interventions: Procedure: Titrated PEEP based on driving pressure
- Conventional (Active Comparator): Conventional PEEP (5cmH2O) is applied.
  Interventions: Procedure: Conventional PEEP

INTERVENTIONS:
Procedure: Titrated PEEP based on driving pressure — Alveolar recruitment and PEEP titration is performed at three time points: after intubation, after Trendelenburg, and after supine after CO2 deflation. The level of PEEP which makes the driving pressure lowest is selected and applied during the operation.
  Arms: Driving pressure
Procedure: Conventional PEEP — Alveolar recruitment is performed at three time points: after intubation, after Trendelenburg, and after supine after CO2 deflation. Conventional PEEP (5cmH2O) is applied during the operation.
  Arms: Conventional

SUMMARY:
The purpose of this study is to investigate the effect of driving-pressure guided positive end-expiratory pressure (PEEP) titration.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robot-assisted laparoscopic prostatectomy with Trendelenburg position

Exclusion Criteria:

* American Society of Anesthesiologists physical status IV or more
* Severe cardiovascular disease
* Severe chronic obstructive pulmonary disease, emphysema
* History of pneumothorax, bullae
* History of lung resection surgery
* Conversion to laparotomy
* Refusal to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Modified lung ultrasound score | 30 minutes after PACU administration
  The score is calculated by adding up the 12 individual part scores assessed using lung ultrasound. The score for each part ranges from 0 to 3.

SECONDARY OUTCOMES:
Modified lung ultrasound score | Intraoperative (at the end of operation before emergence)
  The score is calculated by adding up the 12 individual part scores assessed using lung ultrasound. The score for each part ranges from 0 to 3.
Incidence of intraoperative desaturation | Intraoperative
  Oxygen saturation by pulse oximetry< 95%
Intraoperative partial pressure of arterial oxygen/fraction of inspired oxygen ratio | Intraoperative (30 minutes after designated PEEP applied)
  Partial pressure of arterial oxygen/fraction of inspired oxygen ratio
Postoperative partial pressure of arterial oxygen/fraction of inspired oxygen ratio | 30 minutes after PACU administration
  Partial pressure of arterial oxygen/fraction of inspired oxygen ratio
Postoperative pulmonary complications | After operation~ postoperative day 3
  Extubation failure, Fever, respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, aspiration pneumonitis, pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Susie Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongnogu, South Korea